CLINICAL TRIAL: NCT06607679
Title: Monitoring Intracranial Pressure Change Via Optic Nerve Sheath Ultrasound During Electroconvulsive Therapy
Brief Title: Optic Nerve Sheath Ultrasound During Electroconvulsive Therapy
Status: Completed | Type: Observational
Sponsor: İrem AKSOY (Other)
Collaborators: Cukurova University Medical Faculty Hospital (Unknown)
Responsible Party: Sponsor-Investigator, İrem AKSOY, Consultant Anesthesiologist, Cukurova University
Organization: Cukurova University (Other)
Other Study IDs: 2022-05-03-123/26
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Pressure Change; Hypertension; Electroconvulsive Therapy Treated Patients
Keywords: Intracranial Pressure Change; Hypertension; Electroconvulsive Therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Receiving ECT

SUMMARY:
Electroconvulsive therapy (ECT) is an effective method that has been used for many years in the treatment of psychiatric disorders and is currently administered under general anesthesia. This study evaluated the effect of ECT on intracranial pressure by measuring the optic nerve sheath diameter (ONSD) using ultrasonography. The primary aim was to determine how ONSD values measured during the postictal period change compared to baseline values. Secondary objectives included identifying factors related to the participants and the ECT procedure that affect ONSD.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is a treatment method that has been used effectively for many years in the treatment of psychiatric disorders. Typical uses of ECT include depression, schizophrenia, bipolar disorder, cases resistant to standard therapies, individuals at risk of suicide, and patients exhibiting symptoms of catatonia. The safety of ECT remains a highly debated issue. It is commonly believed that ECT should be avoided in cases of tumors or other space-occupying lesions due to concerns that the therapys stimulus or induced seizure could lead to increased intracranial pressure. The American Psychiatric Association Task Force Report recommends a detailed evaluation of the risk-benefit ratio and measures to minimize the risks associated with the treatment. Measurement of the optic nerve sheath diameter (ONSD) with ultrasound is a direct, noninvasive, and rapid technique for assessing raised ICP. Comparisons between ocular sonography and magnetic resonance imaging (MRI) have shown an acceptable correlation and reliability. In this study, the effects of ECT on intracranial pressure were evaluated by measuring the optic nerve sheath diameter (ONSD) using ultrasonography. The primary aim was to determine the change in ONSD value during the postictal period compared to baseline. Secondary objectives include identifying participants and ECT procedure-related factors affecting ONSD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* ASA 1,2,3
* Participants with various psychiatric problems requiring ECT

Exclusion Criteria:

* Intracranial mass, edema, or bleeding observed on MRI scan
* previous eye surgery
* severe cataracts
* glaucoma
* optic atrophy
* other severe sight impairment
* traumatic brain injury, space-occupying, and inflammatory lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Psychiatry Clinic at the Faculty of Medicine, Cukurova University
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Intracranial Pressure Changes During Electroconvulsive Therapy | 45 MINUTES
  During electroconvulsive therapy, sequential measurements were conducted using ocular ultrasound. These measurements revealed significant changes in intracranial pressure during the post-seizure period compared to baseline values.

SECONDARY OUTCOMES:
Association Between ONSD Measurements And Comorbid Conditions | 45 MINUTES
  An examination of the relationship between increased optic nerve sheath diameter (ONSD) and comorbid conditions revealed that hypertension, higher body mass index, and advanced age were associated with elevated postictal ONSD values.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Laflı Tunay, Associate Professor, Principal Investigator — Department of Anesthesiology and Reanimation, Çukurova University
Locations (1):
- Cukurova University Faculty of Medicine Hospital, Adana, Sariçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I plan to share all IPD that underlie the results in the publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year after publication with no end date.

REFERENCES:
- [Background] Chawla N. Anesthesia for Electroconvulsive Therapy. Anesthesiol Clin. 2020 Mar;38(1):183-195. doi: 10.1016/j.anclin.2019.10.007. Epub 2020 Jan 3. PMID 32008651
- [Background] Singh SK, Bhatia K. Ultrasonographic Optic Nerve Sheath Diameter as a Surrogate Measure of Raised Intracranial Pressure in Severe Pregnancy-induced Hypertension Patients. Anesth Essays Res. 2018 Jan-Mar;12(1):42-46. doi: 10.4103/aer.AER_218_17. PMID 29628552
- [Background] Derikx RL, van Waarde JA, Verwey B, van der Mast RC. Effects on intracranial pressure of electroconvulsive therapy. J ECT. 2012 Jun;28(2):e23-4. doi: 10.1097/YCT.0b013e31824d9b69. PMID 22622301
- [Background] Czosnyka M, Pickard JD. Monitoring and interpretation of intracranial pressure. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):813-21. doi: 10.1136/jnnp.2003.033126. PMID 15145991
- [Background] Bouckaert F, Sienaert P, Obbels J, Dols A, Vandenbulcke M, Stek M, Bolwig T. ECT: its brain enabling effects: a review of electroconvulsive therapy-induced structural brain plasticity. J ECT. 2014 Jun;30(2):143-51. doi: 10.1097/YCT.0000000000000129. PMID 24810772
- [Background] Andrade C, Bolwig TG. Electroconvulsive therapy, hypertensive surge, blood-brain barrier breach, and amnesia: exploring the evidence for a connection. J ECT. 2014 Jun;30(2):160-4. doi: 10.1097/YCT.0000000000000133. PMID 24800688
- [Background] Perera TD, Luber B, Nobler MS, Prudic J, Anderson C, Sackeim HA. Seizure expression during electroconvulsive therapy: relationships with clinical outcome and cognitive side effects. Neuropsychopharmacology. 2004 Apr;29(4):813-25. doi: 10.1038/sj.npp.1300377. PMID 14735129
- [Background] Baghai TC, Moller HJ. Electroconvulsive therapy and its different indications. Dialogues Clin Neurosci. 2008;10(1):105-17. doi: 10.31887/DCNS.2008.10.1/tcbaghai. PMID 18472488
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Background] Andrade C, Arumugham SS, Thirthalli J. Adverse Effects of Electroconvulsive Therapy. Psychiatr Clin North Am. 2016 Sep;39(3):513-30. doi: 10.1016/j.psc.2016.04.004. Epub 2016 Jun 25. PMID 27514303